CLINICAL TRIAL: NCT02269839
Title: A Feasibility Study to Assess the Effectiveness of Different Modalities of Repetitive Transcranial Magnetic Stimulation in the Treatment of Tinnitus
Brief Title: A Feasibility Study Assessing the Effectiveness of rTMS in Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STH15971
Record Dates: First submitted 2014-06-27; First posted 2014-10-21 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Tinnitus
Keywords: Tinnitus; rTMS
MeSH Terms: conditions — Tinnitus | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- theta-burst rTMS (Active Comparator): Active treatment will consist of sessions of continuous theta-burst rTMS on consecutive days for 5 days. This will be delivered with a circular coil to the temporal scalp region overlying the auditory cortex, contralateral to the symptomatic side in unilateral tinnitus and to the left side in bilateral tinnitus. The treatment protocol will consist of treatment at 80% of individual motor threshold (established at the first treatment session) for 600 pulses of 40 seconds duration, which will be repeated after 15 minutes. Each patient will receive 1200 pulses per day.
  Interventions: Device: rTMS
- Control arm (Sham Comparator): The control (sham) stimulation will consist of stimulating with the rTMS coil held at right angles to the participants' head. This will result in no active stimulation of brain tissue but would feel similar to the patient. Each treatment session will therefore last approximately 20 minutes.
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — Active treatment will consist of sessions of continuous theta-burst rTMS on consecutive days for 5 days. This will be delivered with a circular coil to the temporal scalp region overlying the auditory cortex, contralateral to the symptomatic side in unilateral tinnitus and to the left side in bilateral tinnitus. The treatment protocol will consist of treatment at 80% of individual motor threshold (established at the first treatment session) for 600 pulses of 40 seconds duration, which will be repeated after 15 minutes. Each patient will receive 1200 pulses per day.
  Other Names: repetitive Transcranial Magnetic Stimulation

SUMMARY:
Tinnitus is a common problem which can have a severe impact on quality of life and for which there is no truly successful treatment available.

Repetitive transcranial magnetic stimulation (rTMS) is a method of stimulating the brain through the application of a magnetic field in a series of rapid pulses and may be a valuable treatment for patients with tinnitus.

The overall aim of this research is to see if patients with tinnitus benefit from treatment with rTMS, and in particular whether one type (continuous theta burst) is more effective than other variations of rTMS. Prior to developing a definitive study to address this area a feasibility study needs to be performed.

The proposed feasibility study aims to determine outcomes necessary to enable development of a definitive study in the future.

40 patients suffering with idiopathic tinnitus will be randomised into 2 groups, a control group receiving a sham treatment, and an active treatment group receiving theta-burst rTMS on 5 consecutive days.

DETAILED DESCRIPTION:
Tinnitus is a common problem and can have a severe impact on quality of life. At present there is no truly successful treatment available. Repetitive transcranial magnetic stimulation (rTMS) is a method of stimulating the brain through the application of a magnetic field in a series of rapid pulses. Applying it to the areas of the brain thought to be responsible for tinnitus may offer a valuable treatment for patients.

The overall aim of this research is to see if patients with tinnitus benefit from treatment with rTMS, and in particular whether one type (continuous theta burst) is more effective than other variations of rTMS. Prior to developing a definitive study to address this area a feasibility study needs to be performed.

The proposed feasibility study aims to determine outcomes necessary to enable development of a definitive study in the future. Particularly to ensure adequate recruitment will be possible and to confirm the acceptability of the study design to participants. We will assess the success of our chosen placebo intervention and blinding method. The variance in change in tinnitus level following treatment will enable a sample size calculation to be performed for use in future studies.

40 patients suffering with idiopathic tinnitus will be randomised into 2 groups, a control group receiving a sham treatment, and an active treatment group receiving theta-burst rTMS on 5 consecutive days. The effect of treatment will be assessed through the use of the Tinnitus Functional Index an existing validated tinnitus questionnaire. Feasibility outcomes will be assessed through monitoring retention and recruitment rates and the use of questionnaires related to feasibility outcomes

ELIGIBILITY:
Inclusion Criteria:

Age over 18 years

• Persistent unilateral or bilateral subjective tinnitus

Exclusion Criteria:

* Epilepsy

  * Severe or profound hearing loss
  * Patients taking vestibular sedatives, antipsychotic, anxiolytic, antiepileptic and ototoxic medications.
  * Ear infections or discharge
  * History of ear surgery
  * History of noise trauma
  * Excess alcohol consumption
  * Meniere's disease
  * VIII nerve tumour
  * Bells palsy
  * Ramsay-Hunt Syndrome
  * Post-meningitis hearing loss and tinnitus
  * Active psychiatric conditions
  * Congenital or syndromal associations

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Improvement in tinnitus severity following treatment with rTMS | 3 months
  The primary outcome measure for the definitive trial is the improvement in tinnitus severity following treatment with theta burst rTMS compared to control as demonstrated by change in Tinnitus Functional Index (TFI) scores. Assessed on completion of treatment and at 1 week and 1 month following.

SECONDARY OUTCOMES:
The number of patients willing to complete the trial | 3 months
  Feasibility outcome measures relevant to this feasibility study are those which will enable the investigators to successfully complete a full study in the future. One issue is whether sufficient participants could be recruited to run future trials. This will be assessed through measuring the recruitment and retention rate of this feasibility study.
Confirm acceptability of trial design to participants | 3 months
  To enable successful completion of future larger evaluation of patients views on the study design and interventions through simple feedback questionnaires will be performed.
Determine success of sham intervention | 3 months
  To confirm the use and suitability of the control intervention for future trials the investigators will be evaluating whether patients are aware if receiving sham or real rTMS
Success of assessment methods | 3 months
  To evaluate the chosen method and frequency of data collection to evaluate its use for future trials. Assessed by appropriate completion and return of questionnaires.
Sample size calculation | 3 months
  Determination of the number of participants required for a subsequent definitive trial aimed at demonstrating statistical significance.

CONTACTS AND LOCATIONS:
Overall Officials: Jaydip Ray, PhD, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom